CLINICAL TRIAL: NCT00672893
Title: Vibration Response Imaging (VRI) in Patients That Are Undergoing Pulmonary Interventional Procedure
Status: Completed | Type: Observational
Sponsor: Deep Breeze (Industry)
Responsible Party: Prof. Heinrich D. Becker, MD, Thoraxklinik at Heidelberg University
Other Study IDs: DB035-Multi-site; DB020-Single-site
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Central Airway Stenosis
Keywords: central airway stenosis, lung sounds, airway obstruction, bronchial obstruction, bronchoscopic treatment
MeSH Terms: conditions — Respiratory Sounds; Airway Obstruction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients who present to the clinic with airway obstruction and who are designated to undergo intervention
  Interventions: Other: Vibration Response Imaging

INTERVENTIONS:
Other: Vibration Response Imaging — 12 seconds of recording lung sounds

SUMMARY:
Vibration response imaging (VRI) technology, provides a radiation-free dynamic image of the lung, by visualizing vibration energy emitted during the respiration cycle (lung sounds). Airflow in the lungs during the respiration cycle creates vibrations that propagate through the lung tissue; these vibrations are affected by the structural properties of the lungs and may vary in space, time and frequency. Moreover, any structural alteration, such as a bronchial obstruction or space occupying infiltration, is reflected in a corresponding modification of the vibration response.

As obstructions that occur in airways alter airflow, the VRI may provide additional lung function information prior to treatment for airway obstruction and during follow-up. Moreover, the VRI may provide the physician immediate evaluation of the improvement of air flow distribution, quantitative and qualitative measurements. Furthermore, the VRI is a non-invasive, radiation free procedure which is simple and doesn't require the level of patient effort required for lung function test and other evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read and understand the Informed Consent Form and he/she will sign the Informed Consent.
* Male or female in the age range of 18-85 years.
* Body Mass Index >20.
* Patient presented with airway obstruction and who are designated to undergo intervention

Exclusion Criteria:

* Chest wall deformity;
* Spine deformity (including severe scoliosis or kyphosis);
* Hirsutism;
* Potentially contagious skin lesion on the back;
* Skin lesion that would interfere with sensor placement;
* Patient is pregnant;
* Cardiac pacemaker or implantable defibrillator;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the age range of 18-85 and consisting of both male and females, who present to the clinic with airway obstruction and who are designated to undergo intervention.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The principal objective is to determine the ability of the VRI to assess changes in the lungs before and after pulmonary intervention in patients suffering from airway obstruction. | Baseline and follow-up up to 3 months

SECONDARY OUTCOMES:
The secondary objective is to assess the contribution of the VRI in aiding in identification of the pulmonary obstruction as compared to the standard methods prior the intervention procedure. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich D Becker, M.D., Principal Investigator — Thoraxklinik at Heidelberg University School of Medicine
Locations (5):
- United States (2):
  - National Jewish Medical and Research Center, Denver, Colorado
  - Duke University Medical Center, Durham, North Carolina
- Hospital St. Marguerite, Marseille, France
- Thoraxklinik at Heidelberg University, Heidelberg, Germany
- St. Marianna Hospital, Kawasaki, Kanagawa, Japan

REFERENCES:
- [Background] Dellinger RP, Parrillo JE, Kushnir A, Rossi M, Kushnir I. Dynamic visualization of lung sounds with a vibration response device: a case series. Respiration. 2008;75(1):60-72. doi: 10.1159/000103558. Epub 2007 Jun 4. PMID 17551264
- [Background] Ernst A, Feller-Kopman D, Becker HD, Mehta AC. Central airway obstruction. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1278-97. doi: 10.1164/rccm.200210-1181SO. PMID 15187010